CLINICAL TRIAL: NCT02100891
Title: Phase 2 Solid Tumor Immunotherapy Trial Using HLA-Haploidentical Transplant and Donor Natural Killer Cells: The STIR Trial
Brief Title: Phase 2 STIR Trial: Haploidentical Transplant and Donor Natural Killer Cells for Solid Tumors
Acronym: STIR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 15 patients enrolled out of planned 20, terminated due to slow enrollment at end of study
Sponsor: Monica Thakar (Other)
Responsible Party: Sponsor-Investigator, Monica Thakar, Associate Professor of Pediatrics Blood and Marrow Transplant Program, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STIR Trial
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Ewing Sarcoma; Neuroblastoma; Rhabdomyosarcoma; Osteosarcoma; CNS Tumors
Keywords: Ewing Sarcoma; Neuroblastoma; Rhabdomyosarcoma; Osteosarcoma; CNS tumors; Brain Tumors
MeSH Terms: conditions — Sarcoma, Ewing; Neuroblastoma; Rhabdomyosarcoma; Osteosarcoma; Central Nervous System Neoplasms; Brain Neoplasms | interventions — Bone Marrow Transplantation; IL32 protein, human; Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic HCT + Donor NK Cell Infusion (Experimental): Patients will undergo HLA-haploidentical bone marrow transplant preceded by reduced-intensity chemotherapy and radiation therapy, followed by donor NK cells on day +7 after transplant.
  Interventions: Procedure: Allogeneic HCT; Drug: Donor NK Cell Infusion

INTERVENTIONS:
Procedure: Allogeneic HCT — Patients will undergo HLA-haploidentical bone marrow transplant preceded by reduced-intensity chemotherapy and radiation therapy, followed by donor NK cells on day +7 after transplant.
  Other Names: Haplo transplant; Reduced-intensity conditioning; Bone marrow transplant
Drug: Donor NK Cell Infusion — Patients will undergo HLA-haploidentical bone marrow transplant preceded by reduced-intensity chemotherapy and radiation therapy, followed by donor NK cells on day +7 after transplant.
  Other Names: Natural Killer Cells; Adoptive immunotherapy; Donor Lymphocyte Infusion; IND 13794

SUMMARY:
The investigators hypothesize that this Phase 2 cellular and adoptive immunotherapy study using human leukocyte antigen (HLA)-haploidentical hematopoietic cell transplantation (HCT) followed by an early, post-transplant infusion of donor natural killer (NK) cells on Day +7 will not only be well-tolerated in this heavily-treated population (safety), but will also provide a mechanism to treat high-risk solid tumors, leading to improved disease control rate (efficacy). Disease control rate is defined as the combination of complete (CR) and partial (PR) response and stable disease (SD). The investigators further propose that this infusion of donor NK cells will influence the development of particular NK and T cell subtypes which will provide immediate/long-term tumor surveillance, infectious monitoring, and durable engraftment.

Patients with high-risk solid tumors (Ewings Sarcoma, Neuroblastoma and Rhabdomyosarcoma) who have either measurable or unmeasurable disease and have met eligibility will be enrolled on this trial for a goal enrollment of 20 patients over 4 years.

DETAILED DESCRIPTION:
Patients will receive a reduced-intensity conditioning regimen for 6 days that consists of Fludarabine 150 mg/m2, Cyclophosphamide 29 mg/kg, and 3 Gy total body irradiation (TBI), followed by HLA-haploidentical marrow from a family member on Day 0. On Days +3 and +4, Cyclophosphamide 50 mg/kg will be infused for selective in vivo T cell depletion. Additional post-grafting immune suppression will consist of mycophenolate mofetil and either tacrolimus or sirolimus.

Non-mobilized peripheral blood mononuclear cells will be collected from donors on Day +6, from which NK cells will be selected and infused into patients on Day +7.

Patients will be monitored for any transplant-related complications and will undergo disease monitoring every three months for the first two years post-transplant. Research studies will be conducted to follow the patient's immune status and quality of life post-transplant.

ELIGIBILITY:
Inclusion Criteria:

1. No age restrictions
2. Only subjects who are not appropriate candidates for autologous or HLA-matched sibling hematopoietic cell transplants (HCT) may be enrolled.
3. Diseases eligible

   1. High Risk Neuroblastoma (NB): Must have progressed on or recurred after standard frontline therapy including autologous HCT, or be ineligible for autologous HCT.
   2. Ewing Sarcoma Family of Tumors (EWS) [includes both bone and soft tissue Ewing and Peripheral Primitive Neuroectodermal Tumors (PNET)]. Must have progressed on or recurred after standard frontline therapy which includes doxorubicin and ifosfamide.
   3. High-Risk Rhabdomyosarcoma (RMS) or Intermediate Risk Alveolar RMS recurring as more than loco-regional tumor: Must have progressed on or recurred after standard frontline therapy which includes chemotherapy with vincristine, actinomycin, and cyclophosphamide AND either surgery or radiotherapy.
   4. Osteosarcoma: Must have progressed or recurred after standard frontline therapy. If first relapse, must have recurred with a) ≥ 4 lung nodules; b) bilateral lung involvement; or c) relapse outside the lungs.
   5. CNS tumors: High risk malignant brain tumors that are recurrent or refractory to standard frontline therapy are eligible. Diagnoses include: Medulloblastoma, primitive neuro-ectodermal tumor (PNET), ependymoma, high grade (grade 3 or 4) glioma/astrocytoma, germ-cell tumor, or atypical teratoid-rhabdoid tumor (ATRT)

Exclusion Criteria

1. Rapidly-progressing disease prior to HCT, defined as clinical or radiographic evidence of disease progression ≤ 3 weeks prior to protocol registration despite previous achievement of stable or no disease (Appendix C & D) (Note: after disease eligibility has been determined, additional imaging studies are not necessary during the three weeks before the start of conditioning unless there are clinical concerns).
2. Patients who have reached radiation threshold limits and are excluded from receiving 3 Gy TBI.
3. Diffuse intrinsic pontine gliomas (DIPG) are excluded.
4. Performance status: Karnofsky or Lansky <60% Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
5. Patients, who in the opinion of the investigator, may not be able to comply with the treatment plan or safety monitoring requirements of the study Page 16 of 86 Children's Hospital of Wisconsin Medical College of Wisconsin PI: Monica S. Thakar, MD
6. Significant organ dysfunction that would prevent compliance with conditioning, GVHD prophylaxis, or would severely limit the probability of survival, defined as:

   1. Cardiac: For patients not taking inotropic medications and who do not have cardiac failure requiring therapy: Symptomatic coronary artery disease or ejection fraction <35% or, if unable to obtain ejection fraction, shortening fraction of <26%. If shortening fraction is <26% a cardiology consult is required with the PI having final approval of eligibility. For patients taking inotropic medications: Patients displaying corrected cardiac function will be eligible, i.e., patients who take inotropic medications to maintain EF ≥ 35% and SF≥ 26% cardiac function eligibility.
   2. Pulmonary: DLCO <40% TLC <40%, FEV1 <40% and/or receiving supplementary continuous oxygen
   3. Liver: Patient with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension. The patient will be excluded if he/she is found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin >3mg/dL, or symptomatic biliary disease
7. Patients with serious active infections
8. HIV seropositive patients
9. Patients with poorly controlled hypertension despite multiple antihypertensive medications
10. Fertile females who are unwilling to use contraceptive techniques during and for the twelve months following treatment, as well as females who are pregnant or actively breast feeding
11. Fertile males who are unwilling to use contraceptive techniques during and for the twelve months following treatment
12. Life expectancy severely limited by diseases other than malignancy
13. Patients who have received a prior allogeneic HCT are ineligible

DONOR SELECTION An Unrelated Donor Search is not required for entry on this trial. Lack of HLA-matched related or unrelated donors is not a requirement for entry on this trial.

A. Inclusion Criteria

1. Related, HLA-haploidentical donors who are identical for one HLA haplotype and mismatched for any number of HLA-A, -B, -C, DRB1 or DQB1 loci of the unshared haplotype.
2. Marrow will be prioritized as the hematopoietic stem cell source of choice. In cases where adequate stem cells cannot be collected, fresh (preferred) or cryopreserved donor PBSC may be substituted. In the case that PBSC are used, the donor must be 18 years of age or older.
3. HLA-haploidentical donor selection will be based on standard institutional criteria; otherwise no specific prioritization will be made amongst the suitable available donors.

B. Exclusion Criteria

1. Children less than 12 years of age (marrow) or less than 18 years of age (PBSC).
2. Children greater than or equal to 12 years of age who have not provided informed assent in the presence of a parent and an Attending physician who is not a member of the recipient's care team
3. Children greater than or equal to 12-17.9 years of age who have inadequate peripheral vein access to safely undergo apheresis
4. Donors unable or unwilling to undergo marrow harvest or PBSC collection for the initial HCT, storage of autologous blood prior to marrow harvest (if applicable), or apheresis one week after marrow harvest
5. Donors who are not expected to meet the minimum target dose of marrow cells (1 x 108 total nucleated cells/kg recipient weight) for the initial marrow HCT or PBSC transplant (5.0 x 106 CD34/kg recipient weight). The average nucleated cell content of harvested marrow is 22 x 106 nucleated cells/mL or 220 x 108 total nucleated cells/Liter
6. HIV-positive donors
7. Donors who are cross-match positive with recipient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Thakar, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Trial closed early due to low enrollment.
Period: Overall Study
Arm/Group | Allogeneic HCT + Donor NK Cell Infusion
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic HCT + Donor NK Cell Infusion
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 17.2 [4.5 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Disease-control Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic HCT + Donor NK Cell Infusion
Number analyzed (Participants) | 15
Participants | 10

2. Secondary Outcome: Overall Survival
Description: Number of subjects alive at 1 year post-HCT
Time Frame: 1 year
Population: There were 15 subjects enrolled who received the intervention on this 1-armed study.
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic HCT + Donor NK Cell Infusion
Number analyzed (Participants) | 15
Participants | 11

3. Secondary Outcome: Grades 3-4 GVHD
Description: The presence of severe acute grades 3-4 GVHD by day +100
Time Frame: Day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic HCT + Donor NK Cell Infusion
Number analyzed (Participants) | 15
Participants | 0

4. Secondary Outcome: Non-relapse Mortality
Description: Death from causes other than disease by day +100
Time Frame: Day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic HCT + Donor NK Cell Infusion
Number analyzed (Participants) | 15
Participants | 0

5. Secondary Outcome: Progression-free Survival
Description: Alive without progression or relapse of disease by 6 months post-HCT
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic HCT + Donor NK Cell Infusion
Number analyzed (Participants) | 15
Participants | 10

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed up to 1 year post-transplant; all adverse events were collected through 28 days from the NK cell infusion (through day +35 after transplant)
Arm/Group | Allogeneic HCT + Donor NK Cell Infusion
All-Cause Mortality (participants affected / at risk) | 4/15
Serious Adverse Events (participants affected / at risk) | 5/15
Other Adverse Events (participants affected / at risk) | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic HCT + Donor NK Cell Infusion (N=15)
Sepsis (General disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 1 (1)
Febrile neutropenia (General disorders) | 1 (1)
Infection NOS (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic HCT + Donor NK Cell Infusion (N=15)
Fever (General disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to low accrual at end of study leading to lower number of subjects analyzed than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT02100891/Prot_SAP_000.pdf